CLINICAL TRIAL: NCT07153315
Title: Artificial Intelligence-Enhanced Medical Data Analysis for Differentiating Inflammatory and Degenerative Joint Diseases and Detecting of Disease Severity in Elderly Patient
Brief Title: AI-Based Medical Data Analysis for Differentiating Inflammatory vs Degenerative Joint Diseases in Elderly Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Gamea, Principle investigator, Assiut University
Other Study IDs: AU-MEDAI-JOINT-2025-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Arthritis, Rheumatoid (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the diagnostic accuracy of AI-assisted imaging analysis in differentiating between inflammatory and degenerative joint diseases in elderly patients. The performance of AI-based analysis will be compared with radiologists' assessments to determine its reliability in clinical practice. In addition, the study will explore imaging features most predictive of each disease type using advanced machine learning techniques. Finally, the feasibility of implementing AI tools in the routine management of geriatric musculoskeletal disorders will be assessed.

DETAILED DESCRIPTION:
Musculoskeletal disorders are among the most prevalent causes of disability in the elderly. Inflammatory joint diseases, such as rheumatoid arthritis, and degenerative joint diseases, such as osteoarthritis, are both common yet challenging to differentiate, particularly in the early stages. Traditional imaging techniques often lack sensitivity and specificity when interpreted solely by human experts, and diagnostic accuracy is further limited by inter-observer variability.

Artificial Intelligence (AI), particularly deep learning-based image analysis, has emerged as a powerful tool in medical diagnostics. Convolutional neural networks (CNNs), a class of deep learning models, have been successfully applied to musculoskeletal imaging. For example, a study published in The Lancet Rheumatology (2020) trained a CNN on thousands of hand and wrist radiographs from patients with rheumatoid arthritis. The model was able to automatically detect and grade bone erosions and joint space narrowing-key radiographic features of rheumatoid arthritis-with diagnostic performance comparable to experienced musculoskeletal radiologists. Importantly, AI was able to identify early erosive changes in small joints, reduce the time required for radiographic scoring in clinical trials, and provide consistent results, thereby reducing inter-observer variability.

Building on these advances, the current study aims to explore the application of AI in enhancing diagnostic accuracy for differentiating between inflammatory and degenerative joint diseases in elderly patients. By integrating AI-based imaging analysis with clinical and laboratory data, this research will not only support accurate diagnosis but also provide predictive models for disease course, functional decline, and joint damage progression. The ultimate goal is to enable personalized treatment strategies and improve outcomes for elderly patients with musculoskeletal disorders.

ELIGIBILITY:
Inclusion criteria :

1. Age ≥ 60 years
2. Clinical suspicion or confirmed diagnosis of inflammatory joint disease (e.g., rheumatoid arthritis, psoriatic arthritis) or degenerative joint disease (e.g., osteoarthritis)
3. Availability of relevant musculoskeletal imaging (X-rays, MRI, or ultrasound) suitable for AI-based analysis
4. Ability to provide informed consent or have a legal representative consent on behalf of the

Exclusion criteria:

1. History of recent joint trauma (within the last 6 months) or previous joint surgery affecting the studied sites
2. Presence of bone or joint malignancy (primary or metastatic)
3. Diagnosis of overlapping rheumatologic syndromes or mixed pathology (e.g., RA with concurrent gout, or OA with inflammatory overlap)
4. Inadequate imaging quality or absence of required imaging modalities
5. Inability or unwillingness to provide informedconsent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients (≥60 years) presenting to Assiut University Hospitals with clinical suspicion or diagnosis of musculoskeletal disorders, specifically inflammatory joint diseases (such as rheumatoid arthritis) or degenerative joint diseases (such as osteoarthritis), and who have relevant imaging studies (X-ray, MRI, or ultrasound) available for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of AI system | Within 12 months from baseline assessment.
  Sensitivity, specificity, and AUC of AI algorithm for differentiating inflammatory from degenerative joint diseases, using imaging data, compared to expert rheumatologist diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahmoud Mohamed, Resident at internal medicine, Principal Investigator — Assiut University Hospitals - Faculty of Medicine, Assiut University, Egypt
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Bhaumik S. Cardiologists are putting in stents needlessly, doctors say. BMJ. 2013 Feb 4;346:f739. doi: 10.1136/bmj.f739. No abstract available. PMID 23381588
- [Background] Schmidhuber J. Deep learning in neural networks: an overview. Neural Netw. 2015 Jan;61:85-117. doi: 10.1016/j.neunet.2014.09.003. Epub 2014 Oct 13. PMID 25462637
- [Background] Litjens G, Kooi T, Bejnordi BE, Setio AAA, Ciompi F, Ghafoorian M, van der Laak JAWM, van Ginneken B, Sanchez CI. A survey on deep learning in medical image analysis. Med Image Anal. 2017 Dec;42:60-88. doi: 10.1016/j.media.2017.07.005. Epub 2017 Jul 26. PMID 28778026
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39513334/?utm_source=chatgpt.com